CLINICAL TRIAL: NCT06564272
Title: A Phase II Study to Evaluate the Safety and Efficacy of KC1036 in Adolescents Aged 12 and Above With Advanced Ewing Sarcoma
Brief Title: A Study of KC1036 in Adolescents With Advanced Ewing Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Konruns Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC1036-PED-01
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KC1036 (Experimental): oral administration QD
  Interventions: Drug: KC1036

INTERVENTIONS:
Drug: KC1036 — For patients weighing between 30 kg and less than 50 kg, administer 40 mg QD of KC1036. For patients weighing between 50 kg and less than 70 kg, administer 50 mg QD of KC1036. For patients weighing 70 kg or more, administer 60 mg QD of KC1036. 4 weeks as a cycle.

SUMMARY:
This open-label, single-arm clinical trial is to evaluate the safety and effectiveness of KC1036 in treating adolescents aged 12 and above with advanced Ewing sarcoma. Participants will take KC1036 once daily, with each treatment cycle lasting 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and less than 18 years;
* Diagnosed with Ewing sarcoma confirmed by histopathological examination;
* Patients with locally advanced or metastatic Ewing sarcoma that is unresectable or has failed standard treatment, and for whom no other treatment options are available as assessed by the investigator;
* Body weight of ≥30 kg;
* Karnofsky performance status (≥16 years) or Lansky performance status (<16 years) score of ≥60%;
* Patients with at least one measurable lesions according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumors);
* Expected survival of more than 12 weeks;
* Sufficient organ and bone marrow function;
* Female patients who have started menstruating must have a negative pregnancy test;
* The patient and their legal guardians understand and are willing to participate in the trial, and have signed the informed consent form.

Exclusion Criteria:

* Patients with primary central nervous system tumors;
* Presence of central nervous system metastases as diagnosed by imaging;
* History of or concurrent other malignancies within the past 5 years;
* Gastrointestinal abnormalities;
* Cardiovascular or cerebrovascular abnormalities;
* Patients who have previously received VEGFR-TKI small molecule treatment;
* Currently participating in another therapeutic clinical trial; received any anticancer treatment within 2 weeks or 5 half-lives (whichever is longer) before the start of the study treatment; received whole-brain radiation therapy within 14 days before the start of the study treatment; received stereotactic radiosurgery within 7 days before the start of the study treatment; or received herbal or traditional Chinese medicine for anticancer purposes within 2 weeks before the study treatment;
* Underwent major surgery within 2 months before enrollment or have not fully recovered, or plan to undergo surgery during the current study period;
* Persistent toxicity from previous anticancer treatment that has not improved to ≤ Grade 1 (according to CTCAE v5.0), excluding alopecia;
* Unhealed skin wounds, surgical sites, traumatic sites, severe mucosal ulcers, or fractures;
* Uncontrolled significant pleural effusion, ascites, or pericardial effusion;
* Active bacterial, viral, or fungal infections; unexplained fever >38.5°C within 2 weeks before enrollment;
* Hepatitis B surface antigen (HBsAg) positive with HBV-DNA ≥500 IU/mL or 2500 copies/mL; Hepatitis C virus (HCV) antibody positive with HCV RNA ≥200 IU/mL or positive test results; HIV-positive individuals;
* Presence of psychiatric or neurological disorders; or cognitive impairment;
* Fertile patients (e.g., females who have started menstruating or males who have started ejaculating) who do not agree to use contraception (e.g., birth control pills or condoms) during the study and for 6 months after the study ends;
* Patients with insufficient compliance as evaluated by investigator;
* The investigator believes that it is not suitable to patient in this clinical trial.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-27 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | approximately 3 years
  Incidence of treatment-related AEs

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | approximately 3 years
  Overall response rate (ORR) was defined as the percentage of participants with a best overall complete response (CR) or partial response (PR) per RECIST 1.1.
Progression-free survival (PFS) | approximately 3 years
  Progression-free survival (PFS) was defined as the time from the start date of study drug to the date of the first radiologically documented progressive disease (PD) per RECIST 1.1 or death due to any cause.
Disease Control Rate (DCR) | approximately 3 years
  Disease Control Rate (DCR) was defined as the percentage of participants with a best overall complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1.
Duration of Response (DOR) | approximately 3 years
  Duration of response (DOR) was defined as the time from first documented response (partial response (PR) or complete response (CR)) to the date of first documented disease progression (PD) or death due to any cause, among patients with a confirmed PR or CR per RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Huanmin Wang, Principal Investigator — Beijing Children's Hospital Affiliated to Capital Medical University
Locations (1):
- Beijing Children's Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No